CLINICAL TRIAL: NCT01981148
Title: Measurement of Retinal Auto Fluorescence With a Fluorescence Lifetime Imaging Ophthalmoscope
Acronym: FLIO-Group
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: FLIO
Record Dates: First submitted 2013-11-04; First posted 2013-11-11 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Autofluorescence Imaging; Neuroimaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy patients: Healthy patients
  Interventions: Device: Fluorescence lifetime ophthalmoscope
- Patients with various retinal diseases: Various retinal diseases (vascular, hereditary, degenerative)
  Interventions: Device: Fluorescence lifetime ophthalmoscope

INTERVENTIONS:
Device: Fluorescence lifetime ophthalmoscope — All patients and healthy subjects will be imaged with the fluorescence lifetime ophthalmoscope

SUMMARY:
Fluorescent lifetime microscopy has emerged as a useful tool to study fluorescent lifetimes in vitro. Fluorescence lifetime represents the average amount of time a fluorophore remains in the excited state following excitation and depends on the fluorophores molecular environment. Fluorescence lifetime ophthalmoscopy (FLIO) is a technique which can quantify fluorescence lifetimes in the human retina in vivo. The purpose of this study is to investigate fluorescence lifetime characteristics in the human retina by using a FLIO. The investigators hypothesize that FLIO will allow to identify areas of retinal metabolic stress such as ischemia by detecting changes in fluorescence lifetimes.

DETAILED DESCRIPTION:
Background

Ophthalmic imaging has made considerable progress in the last years. Especially the introduction of optical coherence tomography and the scanning laser ophthalmoscope has helped to understand the structural changes underlying various retinal diseases. However, the appearance of structural changes during retinal disease often represents irreversible functional loss with only limited treatment options. In order to prevent loss of vision, retinal diseases should ideally be diagnosed before structural changes occur. This can be achieved by imaging metabolic changes of the retina as most retinal diseases such as age related macular degeneration or diabetic retinopathy are associated with distinct metabolic changes, mainly related to oxidative stress.

Recently, a novel device for imaging fluorescent lifetimes of the retina in vivo, the fluorescent lifetime ophthalmoscope (FLIO), has been developed. This device is able to measure fluorescence lifetimes in the retina on a macroscopic level and may be able to shed new light on metabolic diseases of the retina.

Objective

To define fluorescence lifetime characteristics in healthy patients and patients with various retinal diseases.

Methods

The investigators will use a novel device, the fluorescence lifetime ophthalmoscope (FLIO) to investigate fluorescence lifetimes in the human retina.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be willing to give written informed consent
* Healthy volunteers 18 years of age or greater
* Patients 18 years of age or greater
* No significant media opacities

Exclusion Criteria

* Opacities of ocular media excluding detailed observation of the retina

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients and healthy subjects attending the department of ophthalmology at the University of Bern
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-02; Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Fluorescence lifetime measured by a fluorescence lifetime imaging ophthalmoscope | at baseline
  Measured by fluorescence lifetime variable (TAU). Measured once; in some patients, up to 4 measurements within 2 years will be done

SECONDARY OUTCOMES:
Repeatability of FLIO | at baseline
  Two independent measurements

CONTACTS AND LOCATIONS:
Overall Officials: Martin Zinkernagel, Prof.Dr.Dr., Study Chair — Inselspital, University Clinic Ophthalmology
Locations (1):
- Department of Ophthalmology, Bern University Hospital, Bern, 3010 Bern, Switzerland, Bern, Switzerland

REFERENCES:
- [Result] Klemm M, Dietzel A, Haueisen J, Nagel E, Hammer M, Schweitzer D. Repeatability of autofluorescence lifetime imaging at the human fundus in healthy volunteers. Curr Eye Res. 2013 Jul;38(7):793-801. doi: 10.3109/02713683.2013.779723. Epub 2013 Mar 26. PMID 23530995
- [Result] Schweitzer D, Gaillard ER, Dillon J, Mullins RF, Russell S, Hoffmann B, Peters S, Hammer M, Biskup C. Time-resolved autofluorescence imaging of human donor retina tissue from donors with significant extramacular drusen. Invest Ophthalmol Vis Sci. 2012 Jun 8;53(7):3376-86. doi: 10.1167/iovs.11-8970. PMID 22511622
- [Result] Schweitzer D, Quick S, Klemm M, Hammer M, Jentsch S, Dawczynski J. [Time-resolved autofluorescence in retinal vascular occlusions]. Ophthalmologe. 2010 Dec;107(12):1145-52. doi: 10.1007/s00347-010-2195-7. German. PMID 20552361
- [Result] Dysli C, Quellec G, Abegg M, Menke MN, Wolf-Schnurrbusch U, Kowal J, Blatz J, La Schiazza O, Leichtle AB, Wolf S, Zinkernagel MS. Quantitative analysis of fluorescence lifetime measurements of the macula using the fluorescence lifetime imaging ophthalmoscope in healthy subjects. Invest Ophthalmol Vis Sci. 2014 Apr 3;55(4):2106-13. doi: 10.1167/iovs.13-13627. PMID 24569585
- [Derived] Dysli C, Dysli M, Wolf S, Zinkernagel M. Fluorescence lifetime distribution in phakic and pseudophakic healthy eyes. PLoS One. 2023 Jan 6;18(1):e0279158. doi: 10.1371/journal.pone.0279158. eCollection 2023. PMID 36608033
- [Derived] Lincke JB, Dysli C, Jaggi D, Solberg Y, Wolf S, Zinkernagel MS. LONGITUDINAL FOVEAL FLUORESCENCE LIFETIME CHARACTERISTICS IN GEOGRAPHIC ATROPHY USING FLUORESCENCE LIFETIME IMAGING OPHTHALMOSCOPY. Retina. 2021 Nov 1;41(11):2391-2398. doi: 10.1097/IAE.0000000000003222. PMID 34282069
- [Derived] Dysli C, Dysli M, Lincke J, Jaggi D, Wolf S, Zinkernagel MS. IMAGING ARTIFACTS IN FLUORESCENCE LIFETIME IMAGING OPHTHALMOSCOPY. Retina. 2021 Nov 1;41(11):2378-2390. doi: 10.1097/IAE.0000000000003235. PMID 34111887
- [Derived] Dysli C, Wolf S, Hatz K, Zinkernagel MS. Fluorescence Lifetime Imaging in Stargardt Disease: Potential Marker for Disease Progression. Invest Ophthalmol Vis Sci. 2016 Mar;57(3):832-41. doi: 10.1167/iovs.15-18033. PMID 26934141